CLINICAL TRIAL: NCT07061964
Title: Single Arm Phase II Study of Bladder Preservation With Immunoradiotherapy After a Clinically Meaningful Response to Neoadjuvant Therapy in Patients With Muscle Invasive Bladder Cancer (BRIGHT)
Brief Title: Combining Immunotherapy and Radiation Therapy to Help Patients Avoid Bladder Removal After Treatment Shrinks Muscle Invasive Bladder Cancer, BRIGHT Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2025-04663; NCI-2025-04663 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S2427 (Other: SWOG); S2427 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2025-07-11; First posted 2025-07-14 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Muscle Invasive Bladder Urothelial Carcinoma; Stage II Bladder Cancer AJCC v8; Stage IIIA Bladder Cancer AJCC v8
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Specimen Handling; Cystoscopy; Magnetic Resonance Spectroscopy; pembrolizumab; Photons; Radiation; Transurethral Resection of Bladder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (photon beam RT, pembrolizumab) (Experimental): Patients undergo photon beam RT QD on Monday-Friday for up to 20 treatments and receive pembrolizumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 21 days for up to 18 cycles (for a total of 12 months, including NAT) in the absence of disease progression or unacceptable toxicity. Patients also undergo TURBT with tissue sample collection at pre-registration and CT, MRI or PET, cystoscopy, and urine and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Cystoscopy; Procedure: Magnetic Resonance Imaging; Biological: Pembrolizumab; Radiation: Photon Beam Radiation Therapy; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Procedure: Transurethral Resection of Bladder Tumor

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo tissue, urine, and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Cystoscopy — Undergo cystoscopy
  Other Names: CS
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475
Radiation: Photon Beam Radiation Therapy — Undergo photon beam RT
  Other Names: External beam radiation therapy using photons (procedure); Photon; Photon EBRT; Photon External Beam Radiotherapy; PHOTON Therapy; Radiation, Photon Beam
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Other: Questionnaire Administration — Ancillary studies
Procedure: Transurethral Resection of Bladder Tumor — Undergo TURBT
  Other Names: Transurethral resection (TURBT); TURBT

SUMMARY:
This phase II trial tests the effect of giving pembrolizumab in combination with radiation therapy after chemotherapy in preventing surgery to remove the bladder in patients with muscle invasive bladder cancer. Standard of care therapy includes chemotherapy before surgery (neoadjuvant) to shrink or get rid of the tumor. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the tumor, and may interfere with the ability of tumor cells to grow and spread. Radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill cancer cells and shrink tumors. Photon beam radiation therapy is a type of radiation therapy that uses x-rays or gamma rays that come from a special machine called a linear accelerator. The radiation dose is delivered at the surface of the body and goes into the tumor and through the body. Giving pembrolizumab in combination with radiation therapy after neoadjuvant chemotherapy may help prevent surgical removal of the bladder in patients with muscle invasive bladder cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate whether 3-year bladder intact event-free survival (BI-EFS) is at least 70% in participants with clinically T0-clinically T1 without multifocal carcinoma in situ (CIS) following neoadjuvant therapy (NAT) for muscle-invasive bladder cancer (MIBC) who receive radiotherapy (RT) + pembrolizumab (MK-3475).

SECONDARY OBJECTIVES:

I. To estimate BI-EFS in participants who receive RT + pembrolizumab (MK-3475). II. To estimate local muscle invasive recurrence-free survival in participants who receive RT+ pembrolizumab (MK-3475).

III. To estimate the metastasis-free survival (MFS) in participants who receive RT+ pembrolizumab (MK-3475).

IV. To estimate the overall survival (OS) in participants who receive RT + pembrolizumab (MK-3475).

V. To estimate the rate of salvage cystectomy in participants who receive RT+ pembrolizumab (MK-3475).

VI. To evaluate the frequency and severity of toxicities in participants who receive RT + pembrolizumab (MK-3475).

PATIENT REPORTED OUTCOMES (PRO)-COMMON TERMINOLOGY CRITERIA FOR ADVERSE EVENTS (CTCAE) OBJECTIVE:

I. To evaluate participant-reported symptoms using selected items from Gastrointestinal, Genitourinary and sexual function domains of the PRO-CTCAE, with the goal of characterizing the frequency, severity, and interference of treatment-related symptoms.

BANKING OBJECTIVE:

I. To bank specimens for future correlative studies.

OUTLINE:

Patients undergo photon beam RT once daily (QD) on Monday-Friday for up to 20 treatments and receive pembrolizumab intravenously (IV) over 30 minutes on day 1 of each cycle. Cycles repeat every 21 days for up to 18 cycles (for a total of 12 months, including NAT) in the absence of disease progression or unacceptable toxicity. Patients also undergo transurethral resection of bladder tumor (TURBT) with tissue sample collection at pre-registration and computed tomography (CT), magnetic resonance imaging (MRI) or positron emission tomography (PET), cystoscopy, and urine and blood sample collection throughout the study.

After completion of study treatment, patients are followed every 26 weeks until year 2 and then every 52 weeks up to year 5.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologic evidence of cT2-T4aN0M0 muscle invasive urothelial carcinoma of the bladder within 180 days prior to starting neoadjuvant therapy (NAT)
* Participants must have had CT chest/abdomen/pelvis (C/A/P), MRI C/A/P or PET within 60 days prior to starting NAT to determine cT2-T4aN0M0
* Participants must have undergone TURBT with biopsy of areas of prior disease and systematic biopsies (left and right lateral, dome, posterior wall and trigone) and radiologic staging showing clinically T0-T1 disease within 60 days after the last dose of NAT. At least 4 out of 5 systematic biopsies must be performed

  * NOTE: This TURBT must be within 90 days prior to registration. Registration must be within 90 days after the last dose of NAT
* Participants must have imaging of the chest, abdomen, and pelvis performed using CT or MRI preferably with contrast. Fludeoxyglucose F-18 (FDG) PET-CT can also be used for staging. If FDG PET-CT is used, then it is at the discretion of the investigator if they want to additionally obtain diagnostic CT or MRI with contrast within 60 days after the last dose of NAT
* Participants with lymph nodes ≥ 1.0 cm in the shortest cross-sectional diameter on imaging (CT or MRI of abdomen and pelvis) after completion of NAT must have a PET-CT within 70 days prior to registration. A biopsy in the setting of negative PET-CT is not required unless there is strong clinical suspicion for nodal involvement with tumor. Participants with a positive PET are deemed ineligible unless a biopsy is performed and shows no evidence of tumor involvement

  * NOTE: For questions regarding the above eligibility criteria, please contact the study chairs in addition to the Southwest Oncology Group (SWOG) Statistics and Data Management Center (SDMC)
* Participants must not have evidence of ≥ T2, or N1-3, or M1 disease after NAT
* Participants must not have the presence of small cell, neuroendocrine carcinoma, plasmacytoid variants on any pathology
* Participants must not have had urothelial carcinoma or histological variant at any site outside of the urinary bladder within 24 months prior to registration except Ta/T1/carcinoma in situ (CIS) of the upper urinary tract, including renal pelvis or ureter if the participant underwent complete nephroureterectomy

  * NOTE: Participants with mixed variant histology will be eligible for the trial if the majority (> 50%) of the tumor is urothelial cell carcinoma
* Participants will be allowed to continue PD-1/L-1 inhibitor therapy received as part of standard of care neoadjuvant therapy while they undergo pre-registration assessments (TURBT and imaging)
* Participants must have received at least 3 and no more than 6 cycles of Food and Drug Administration (FDA) approved NAT for MIBC. These include cisplatin-based combination chemotherapy (e.g. cisplatin and gemcitabine [GC] with or without PD-1/L1 inhibitors) dose dense or accelerated methotrexate, vinblastine, doxorubicin and cisplatin (MVAC) or enfortumab vedotin with PD-1/L1 inhibitor
* Participants must not have had anti-PD-1, anti PD-L1, anti PD-L2 or anti-CTLA4 antibody, any other antibody or drug targeting T-cell co-stimulation, enfortumab vedotin, or any other drug targeting nectin-4 other than for neoadjuvant treatment for MIBC

  * NOTE: Prior intravesical immunotherapy or chemotherapy for non-muscle invasive disease is allowed
* Participants must not have had prior pelvic radiotherapy
* Participants must not have received a live attenuated vaccination within 28 days prior to registration
* Participants with conditions requiring immunosuppressive doses of steroids (> 10 mg/day of prednisone or equivalent) or other immunosuppressive medications must not be taking steroids at time of trial registration
* Participants must be ≥ 18 years old at the time of registration
* Participants must have Zubrod performance status of 0-2
* Participants must have a complete medical history and physical exam within 28 days prior to registration
* Leukocytes ≥ 3 x 10^3/uL (within 28 days prior to registration)
* Absolute neutrophil count ≥ 1.5 x 10^3/uL (within 28 days prior to registration)
* Platelets ≥ 100 x 10^3/uL (within 28 days prior to registration)
* Total bilirubin ≤ institutional upper limit of normal (ULN) unless history of Gilbert's disease (within 28 days prior to registration)

  * Participants with history of Gilbert's disease must have total bilirubin ≤ 5 x institutional ULN
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 3 x institutional ULN (within 28 days prior to registration)
* Participants must have a creatinine ≤ the institutional (I)ULN OR measured OR calculated creatinine clearance ≥ 40 mL/min using the following Cockcroft-Gault Formula. This specimen must have been drawn and processed within 28 days prior to registration
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class II or better
* Participants with a history of human immunodeficiency virus (HIV)-infection must be on effective anti-retroviral therapy at registration and have undetectable viral load test on the most recent test results obtained within 6 months prior to registration
* For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured (defined as undetectable HCV viral load)
* Participants must not have a prior or concurrent malignancy whose natural history or treatment (in the opinion of the treating physician) has the potential to interfere with the safety or efficacy assessment of the investigational regimen
* Participants must not be pregnant or nursing (nursing includes breast milk fed to an infant by any means, including from the breast, milk expressed by hand, or pumped). Individuals who are of reproductive potential must have agreed to use an effective contraceptive method with details provided as a part of the consent process. A person who has had menses at any time in the preceding 12 consecutive months or who has semen likely to contain sperm is considered to be of "reproductive potential." In addition to routine contraceptive methods, "effective contraception" also includes refraining from sexual activity that might result in pregnancy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) including hysterectomy, bilateral oophorectomy, bilateral tubal ligation/occlusion, and vasectomy with testing showing no sperm in the semen
* Participants must be offered the opportunity to participate in specimen banking
* Participants who can complete the PRO-CTCAE questionnaire in English or Spanish will be offered the opportunity to participate in the optional patient-reported outcome study
* NOTE: As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

  * Participants must be informed of the investigational nature of this study and must sign and give informed consent in accordance with institutional and federal guidelines
  * For participants with impaired decision-making capabilities, legally authorized representatives may sign and give informed consent on behalf of study participants in accordance with applicable federal, local, and central institutional review board (CIRB) regulations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Bladder intact event-free survival (BI-EFS) | Within 3 years after registration
  Will be evaluated as the percentage of participants who do not experience a BI-EFS event using a Kaplan-Meier estimate. A single-arm test of proportions will be used to test against the null hypothesis (true BI-EFS = 55%). Standard errors will be calculated using Greenwood's formula. If the upper bound of the one-sided 90% confidence interval includes 70%, then the radiation therapy + pembrolizumab regimen will be concluded to be active in this population.

SECONDARY OUTCOMES:
BI-EFS | From registration to the first documentation of a BI-EFS event, assessed up to 5 years
Local muscle invasive recurrence-free survival | From date of registration to first radiologic or histologic evidence of local muscle invasive bladder carcinoma recurrence, assessed up to 5 years
Metastasis-free survival | From date of registration to first radiologic or histologic evidence of metastatic disease or death due to any cause, assessed up to 5 years
Overall survival | From date of registration to date of death due to any cause, assessed up to 5 years
Salvage cystectomy | Up to 5 years
  Will be defined as the number of participants that undergo a radical cystectomy.
Incidence of adverse events | Up to 30 days after last dose of study treatment
  Will be assessed using National Cancer Institute CTCAE version 5.0.

OTHER OUTCOMES:
Patient reported adverse events | Up to 5 years
  Selected Patient Reported Outcomes (PRO)-Common Terminology Criteria for Adverse Events (CTCAE) questions will be used to assess patient-reported symptoms. For each of the PRO-CTCAE adverse events examined, the scores for each attribute (frequency, severity and/or interference) will be presented descriptively using summary statistics at each assessment time. Additionally, the worst level of frequency, severity and/or interference over the entire course will be summarized. The proportion of patients by arm experiencing a maximum follow-up PRO-CTCAE score greater than 0 (reflecting any evidence of a given symptom) or 3 or higher (reflecting "frequent" or worse, "severe" or worse, or "quite a bit" or worse of frequency, severity, and interference items, respectively), both unadjusted and adjusted for the baseline PRO-CTCAE score, will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Ballas, Principal Investigator — SWOG Cancer Research Network
Locations (111):
- United States (111):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Tower Cancer Research Foundation, Beverly Hills, California
  - City of Hope Corona, Corona, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope at Irvine Lennar, Irvine, California
  - City of Hope Antelope Valley, Lancaster, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - City of Hope South Pasadena, South Pasadena, California
  - Cedars-Sinai Cancer - Tarzana, Tarzana, California
  - City of Hope Upland, Upland, California
  - Shaw Cancer Center, Edwards, Colorado
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Moffitt Cancer Center at SouthShore, Ruskin, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Moffitt Cancer Center at Wesley Chapel, Wesley Chapel, Florida
  - CTCA at Southeastern Regional Medical Center, Newnan, Georgia
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Northwestern Medicine Oak Brook, Oak Brook, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - The Iowa Clinic PC, West Des Moines, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Fairview Southdale Hospital, Edina, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Community Medical Center, Missoula, Montana
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - UT Southwestern Simmons Cancer Center - RedBird, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm